CLINICAL TRIAL: NCT05073900
Title: Comparison of the Efficacy of Ultrasound Guided Rhomboid Intercostal Block and Erector Spinal Plane Block on Lower Cervical and Interscapular Myofascial Pain Syndrome
Brief Title: Comparison of the Efficacy of Rhomboid Intercostal Block and Erector Spinal Plane Block on Myofascial Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, Selin Guven Kose, Principal Investigator, Diskapi Teaching and Research Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 107/29
Record Dates: First submitted 2021-09-29; First posted 2021-10-12 (Actual); Last update posted 2021-11-29 (Actual); Status verified 2021-11

CONDITIONS: Myofascial Pain Syndrome
MeSH Terms: conditions — Myofascial Pain Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rhomboid intercostal block (Experimental): Ultrasound guided rhomboid intercostal block
  Interventions: Procedure: Rhomboid intercostal block
- Erector spinae plane block (Active Comparator): Ultrasound guided erector spinae plane block
  Interventions: Procedure: Rhomboid intercostal block

INTERVENTIONS:
Procedure: Rhomboid intercostal block — two regional anesthesia block techniques are applied
  Other Names: Erector spinae plane block

SUMMARY:
The investigators evaluate the effect of Ultrasound guided Rhomboid Intercostal Block and Erector Spinal Plane Block on lower cervical and inter scapular Myofascial Pain

DETAILED DESCRIPTION:
Myofascial pain syndrome (MPS) is the most common cause of musculoskeletal pain and its prevalence in the population is reported to be 21-30%. In this study, the investigators compare the effect of two regional anesthesia block techniques with the ultrasound guidance.

ELIGIBILITY:
Inclusion Criteria:

* Complaint of myofascial pain
* Pain that is rated at least 3 on a numerical rating scale (NRS, 0 = no pain, 10 = the worst pain)

Exclusion Criteria:

* pregnancy
* presence of coagulopathy, or the use of anticoagulants
* a history of surgery on the block area
* allergic to bupivacaine
* decline to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-07-10 (Actual); Primary Completion 2021-09-10 (Actual); Study Completion 2021-10-24 (Actual)

PRIMARY OUTCOMES:
Numerical Rating Scale (NRS) | Change from baseline to minutes 30, day 1, week 1, 2, 4, 6 after the block
  Pain Score Change The 11-point NRS consists of numbers between 0 and 10 where 0 indicates "no pain" and 10 indicates "maximum pain." The patient is instructed to identify one number between 0 and 10, which is best representative of their pain intensity.

CONTACTS AND LOCATIONS:
Overall Officials: selin guven kose, Principal Investigator — Diskapi Teaching and Research Hospital
Locations (1):
- Diskapi Yildirim Beyazit Training and Research Hospital, Ankara, Turkey (Türkiye)